CLINICAL TRIAL: NCT04379869
Title: A Combined Single Dose and Multiple Ascending Dose Study to Assess the Safety, Tolerability and Pharmacokinetic Profile of NNZ-2591 in Healthy Volunteers
Brief Title: To Evaluate the Safety, Tolerability and Pharmacokinetics of Oral NNZ-2591 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuren Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NEU-2591-HV-001
Record Dates: First submitted 2020-04-30; First posted 2020-05-08 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers
MeSH Terms: interventions — cyclo-L-glycyl-L-2-allylproline

STUDY DESIGN:
Intervention Model Description: Stage 1: Open-label, single dose with 2 dose cohorts. Stage 2: Randomised, Double-blind, Placebo-controlled, Multiple Ascending Dose (MAD) with 2 dose cohorts
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stage 1: None Stage 2: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NNZ-2591 Single dose Cohort 1 (Experimental): Single dose of oral NNZ-2591 in healthy volunteers
  Interventions: Drug: NNZ-2591
- NNZ-2591 Single dose Cohort 2 (Experimental): Single dose of oral NNZ-2591 in healthy volunteers
  Interventions: Drug: NNZ-2591
- NNZ-2591 MAD Cohort 1 (Experimental): Multiple Ascending Dose (MAD) of oral NNZ-2591 in healthy volunteers
  Interventions: Drug: NNZ-2591; Drug: Placebo
- NNZ-2591 MAD Cohort 2 (Experimental): Multiple Ascending Dose (MAD) of oral NNZ-2591 in healthy volunteers
  Interventions: Drug: NNZ-2591; Drug: Placebo

INTERVENTIONS:
Drug: NNZ-2591 — Single dose of NNZ-2591
Drug: Placebo — Comparator for double-blind MAD
  Arms: NNZ-2591 MAD Cohort 1; NNZ-2591 MAD Cohort 2

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of NNZ-2591 when administered to healthy volunteers.

DETAILED DESCRIPTION:
This study is in two stages:

Stage 1: A First-in-Human (FIH), single dose escalation study of oral NNZ-2591 in healthy volunteers to establish safety, tolerability and pharmacokinetic parameters.

Stage 2: A First-in-Human (FIH), randomised, double-blind, placebo-controlled, Multiple Ascending Dose study (MAD) in healthy volunteers to establish safety, tolerability and pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 55 years, inclusive;
2. Weight at screening and admission between 45 kg and 100 kg;
3. Body mass index (BMI) between 18.0 and 32.0 kg/m2 inclusive;
4. Healthy as determined by the Investigator based on pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead electrocardiogram (ECG);
5. Negative tests for Hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV) and human immunodeficiency virus (HIV)-1 and HIV-2 antibody at screening;
6. Clinical laboratory test results up to >1.5 x Lower Limit of Normal (LLN) or <1.5 x Upper Limit of Normal (ULN) at screening and admission and deemed not clinically significant by the Investigator;
7. Negative screen for alcohol and drugs of abuse at screening and admission;
8. Non-smokers or ex-smokers (must have ceased smoking >3 months prior to screening visit);

   If female:
9. Woman with no childbearing potential by reason of surgery or at least 1year post- menopause (i.e., 12 months post last menstrual period), and menopause confirmed by follicle-stimulating hormone (FSH) testing;
10. If of childbearing potential, using an effective nonhormonal method of contraception (intrauterine device; condom or occlusive cap [diaphragm or cervical or vault caps]; true abstinence; or vasectomized male partner (provided that he is the sole partner of that subject and had a vasectomy ≥30 days prior to screening) for the duration of the study and up to one month after the last investigational medicinal product (IMP) administration;
11. Negative serum pregnancy test at screening and negative urine pregnancy test on admission (women of childbearing potential only);

    If male:
12. Using an effective method of contraception (condom) if sexually active with a female partner of child-bearing potential; true abstinence; or vasectomy ≥30 days prior to screening) throughout the study and for one month after the last IMP administration.

Exclusion Criteria:

1. Subjects who have a clinically relevant history as determined by the Investigator, or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders;
2. Fridericia's correction factor for QT (QTcF) > 450 ms for male participants and >470ms for female participants or history of QT interval prolongation.
3. Have a clinically relevant surgical history, as determined by the Investigator;
4. Have a history of relevant atopy or drug hypersensitivity;
5. Have a history of alcoholism or drug abuse;
6. Consume more than 21 standard drinks a week for males and more than 14 standard drink if female [1 standard drink is any drink containing 10g of alcohol, regardless of container size or alcohol type].
7. Have a significant infection or known inflammatory process on screening or admission;
8. Have acute gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea, heartburn) at the time of screening or admission;
9. Have used any prescription or non-prescription medicines within 2 weeks of admission, unless in the investigator's opinion will not affect determination of safety or other study assessments. Occasional paracetamol use (up to 2g/day is permitted);
10. Have received any investigational drug within 30 days prior to screening;
11. Have used tobacco or nicotine products within 3 months of screening
12. Have donated or received any blood or blood products within the 3 months prior to screening;
13. Cannot communicate reliably with the investigator;
14. Are unlikely to co-operate with the requirements of the study;
15. Are unwilling or unable to give written informed consent.

    If female:
16. Pregnancy or breast-feeding;
17. Woman of childbearing potential not willing to use an accepted effective contraceptive method or using hormonal contraceptives;

    If male:
18. Not willing to use an accepted effective method of contraception.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability measured through Adverse Events /Serious Adverse Events | 25 days
  The frequency and severity of Adverse Events in healthy volunteers administered single and repeated oral doses of NNZ-2591

SECONDARY OUTCOMES:
Pharmacokinetic - Cmax | 17 days
  Maximum observed plasma concentration (Cmax) of NNZ-2591
Pharmacokinetic - AUC∞ | 17 days
  Area under the concentration-time curve from time 0 to infinity of NNZ-2591
Pharmacokinetic - Tmax | 17 days
  Time to Cmax of NNZ-2591
Pharmacokinetic - t1/2 | 17 days
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: James Shaw, Study Director — Neuren Pharmaceuticals; Jasmine Williams, Principal Investigator — Linear Clinical Research
Locations (2):
- Australia (2):
  - Scientia Clinical Research, Sydney, New South Wales
  - Linear Clinical Research, The Queen Elizabeth II Medical Centre, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No